CLINICAL TRIAL: NCT06415955
Title: Identification of Limiting Factors in the Locomotor Activity of Individuals With Lower Limb Amputation: Biomechanical, Physiological, Psychological.
Brief Title: Identification of Limiting Factors in the Locomotor Activity of Individuals With Lower Limb Amputation:
Acronym: AMPUTEEFACT
Status: Not yet recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: LOCAL/2024/EP-01; IRB 24.03.08 (Other: IRB CHU de Nîmes)
Record Dates: First submitted 2024-05-13; First posted 2024-05-16 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Lower Limb Amputation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Lower Limb Amputation: Patients with lower limb amputations, unilateral or bilateral, walking with or without technical aids, at any level (trans-femoral or trans-tibial) and hospitalised in the locomotor rehabilitation department of the Nîmes University Hospital.
  Interventions: Other: None, pure observationnal study

INTERVENTIONS:
Other: None, pure observationnal study — None, pure observationnal study

SUMMARY:
The experience of amputation leads to a deterioration in quality of life, with undeniable somatic and functional repercussions. The result is a reduction in general mobility, increased metabolic energy requirements and a feeling of discomfort and pain. The rehabilitation objectives focus on improving, or at least maintaining, the range of movement of the lower limbs, strengthening the overall muscles, ensuring that the equipment is correctly adapted, re-training for physical exertion and working on balance and walking. The rehabilitation objectives focus on social inclusion with the equipment, to optimise the return home and promote social and professional reintegration, and therapeutic education. Factors influencing the postoperative resumption of walking in amputees have been identified as key elements in the success of rehabilitation management. These include maintaining joint range of motion before fitting any equipment, combating postoperative loss of muscle mass, managing cardiorespiratory deconditioning and, finally, resuming walking with the aid of equipment, taking account of fluctuating balance.

The literature shows that a change in the centre of gravity and postural instability, particularly when changing stance, are responsible for a greater risk of falls in lower-limb amputees. This asymmetry of gait, which is the cause of a greater risk of secondary joint degeneration, is found in both transtibial and transfemoral amputees. This alteration in balance has a direct influence on walking ability, and therefore calls for significant proprioceptive management in the rehabilitation programme. Gait analysis in lower-limb amputees therefore seems essential, both for the purposes of evaluating and monitoring rehabilitation treatment, and for prosthetic selection and adjustment. Three-dimensional assessment of walking in amputees, coupled with force platforms, is the test of choice for providing kinematic, kinetic and spatiotemporal data (motion capture).

ELIGIBILITY:
Inclusion Criteria:

* Amputees in PRM hospitalisation at the CHU Nîmes RRL service University Rehabilitation Hospital in Le Grau du Roi.
* All aetiologies: vascular, traumatic and septic.
* Appropriate vascular equipment validated by PRM doctor.
* Able to walk for 5 minutes on a treadmill.
* Patient affiliated to or benefiting from a health insurance scheme.
* Adult patient (>18 years) and under 80 years of age.

Exclusion Criteria:

* Patients with uncorrected or untreated visual disorders.
* Patients with major cognitive impairment (MOCA>23).
* Patients with vestibular disorders.
* Patient with uncontrolled epilepsy.
* Patient with an unhealed amputation stump.
* Weight > 135kg or < 20kg
* Patients with a FAC of 1 (i.e. patients requiring the firm and continuous assistance of another person to carry their weight and maintain their balance) or less.
* Inability to properly adjust the sling to the corresponding body part due to:
* Body shape
* Colostomy bags
* Skin lesions that cannot be adequately protected.
* Any other reason that prevents the harness from being adjusted correctly and painlessly.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with lower limb amputations, unilateral or bilateral, walking with or without technical aids, whatever the level (trans-femoral or trans-tibial) and hospitalised in the locomotor rehabilitation department. Patients who were not autonomous enough to walk and required a third person (human aid) were not included.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
VO2 consumption as a function of amputation level | Before and during performance of a standardised motor task
  To quantify the cost (consumption of Vo2 in mL/kg/min) of a task as a function of the level of amputation. VO2 consumption is measured using a VO2 master calorimetric mask, which analyses gas exchange for 3 minutes. To quantify the cost of the task, VO2 consumption over the 3rd minute is used, normalised in relation to VO2 consumption at rest.
VO2 consumption as a function of gait asymmetry | Before and during performance of a standardised motor task
  Quantify the cost (Vo2 consumption in mL/kg/min) of a task as a function of gait asymmetry compared with VO2 consumption at rest.
Consumption of VO2 as a function of prosthetic equipment | Before and during performance of a standardised motor task
  To quantify the cost (consumption of Vo2 in mL/kg/min) of a task as a function of the prosthetic equipment compared with the consumption of VO2 at rest.
Consumption of VO2 as a function of walking condition. | Before and during performance of a standardised motor task
  To quantify the cost (consumption of Vo2 in mL/kg/min) of a task as a function of the walking condition compared with the consumption of VO2 at rest.

CONTACTS AND LOCATIONS:
Overall Officials: Anissa MEGZARI, Study Director — Centre Hospitalier Universitaire de Nīmes